CLINICAL TRIAL: NCT05190679
Title: Prospective Phenotyping for Genetic Subtypes of Early-onset Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, M. Benjamin Shoemaker, Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 210819; R01HL155197 (NIH)
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: Genetic disease
MeSH Terms: conditions — Atrial Fibrillation; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Whole blood samples retained for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiomyopathy Rare Variant Cases: Identified Pathogenic/Likely pathogenic rare variant in cardiomyopathy (CM) gene which include inherited CM syndromes.
  Interventions: Other: None/Observational Studies
- Arrhythmia Rare Variant Cases: Identified Pathogenic/Likely pathogenic rare variant in arrhythmia genes.
  Interventions: Other: None/Observational Studies
- Controls: No rare variant in CM, arrhythmia, or other atrial fibrillation gene.
  Interventions: Other: None/Observational Studies

INTERVENTIONS:
Other: None/Observational Studies — This is an observational study and there is no intervention.

SUMMARY:
This is a prospective, case-control study that seeks to learn about the role of genetics in early onset atrial fibrillation (AF) and if genetic testing can be used to improve how the investigators treat atrial fibrillation. The study will enroll 225 participants. Eligible participants will have undergone sequencing for arrhythmia and cardiomyopathy (CM) genes. Based on those results, participants will be recruited for an outpatient research visit with testing that includes cardiac MRI, rest/stress/signal-averaged ECGs, and cardiac monitoring. If an inherited arrhythmia/CM syndrome is diagnosed, guideline-directed changes to medical care will be recommended.

DETAILED DESCRIPTION:
This study will address the hypothesis that re-phenotyping patients with AF and pathogenic arrhythmia/CM variants will identify unrecognized underlying genetic disease.

The investigators will recruit from participants sequenced as part of our prospective clinical registries and participants cared for in the Vanderbilt Genetic Arrhythmia Clinic or Meharry Arrhythmia Clinic and enrolled in the Vanderbilt Early-onset Atrial Fibrillation Registry (IRB #201666). Eligible participants will have pathogenic/likely pathogenic (P/LP) rare variants (or matched controls) and will undergo prospective cardiac phenotyping, which will include a cardiac MRI, rest/stress/signal averaged ECGs, blood work, and ambulatory ECG monitoring. A subset of patients will also undergo a procainamide drug challenge. If an inherited arrhythmia/CM syndrome is diagnosed, guideline-directed changes to medical care will be recommended.

This study will define the cardiac phenotype of individuals with AF who have a P/LP rare variant in an inherited arrhythmia or CM disease gene and compare to controls. Participants with a P/LP variant in a cardiomyopathy gene or arrhythmia gene (N=150) will be compared to controls (N=75). Controls will have no P/LP variant and be balanced for sex, race, and ethnicity. The association between P/LP variants and the following endpoints will be tested: 1) imaging and ECG-derived measurements (e.g., ventricular size, function, fibrosis, ectopy); 2) diagnoses (e.g., arrhythmogenic cardiomyopathy (AC), hypertrophic cardiomyopathy (HCM), dilated cardiomyopathy (DCM), Long QT Syndrome (LQTS), Short QT Syndrome (SQTS), Brugada Syndrome, Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT), Progressive Cardiac Conduction Disease (PCCD); and 3) management changes including new medical therapy, activity restrictions, implantable cardioverter-defibrillator use, or cascade screening. Sample sizes per group have been selected to power the diagnostic and management endpoints. An Adjudication Committee with arrhythmia, CM, and genetics expertise will determine if diagnostic criteria are met and make management recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Minors >15 years
* Adult > 18 years
* Able to provide written informed consent
* Previously enrolled in the Vanderbilt Atrial Fibrillation Registry (IVR#020669)
* Atrial Fibrillation Ablation Registry (IRB#110881)
* Early-onset Atrial Fibrillation Registry (IRB#201666)
* Underwent whole genome sequencing/whole exome sequencing or clinical genetic testing and based on those results meets the genetic criteria for cases and controls as defined as a Cardiomyopathy (CM) Rare Variant (P/LP rare variant in CM gene, Arrhythmia Rare Variant (P/LP rare variant in arrhythmia gene), or a Control (no rare variant in CM, arrhythmia, or other Atrial Fibrillation gene).
* Diagnosis of Atrial Fibrillation prior to age of 65 (</=65)

Exclusion Criteria:

-Pregnant women

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Previous participants who were enrolled in the Vanderbilt Atrial Fibrillation Registry (IVR#020669), Atrial Fibrillation Ablation Registry (IRB#110881), or Early-onset Atrial Fibrillation Registry (IRB#201666).
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Inherited Cardiomyopathy (CM) Syndromes. | 6 weeks
  Clinical data and results are reviewed by the Adjudication Committee to determine if criteria for diagnostic endpoints are met for each participant that has completed the phenotyping protocol. The committee will remain blinded to the participant's genotype until the discussion of the clinical phenotyping result has ended. Genetic test results will be revealed and final determination of the diagnosis will be made. The Adjudication Committee will use published diagnostic criteria for specific inherited CM syndromes: Arrhythmogenic cardiomyopathy (AC), Arrhythmogenic Right Ventricular CM (ARVC), Dilated CM (DCM), Hypertrophic CM (HCM), and Left Ventricular Noncompaction CM (LVNC). For AC and DCM, only participants determined to have "definite" AC or DCM according to the diagnostic criteria will be considered as meeting the primary diagnostic endpoint.
Number of Participants with Inherited Arrhythmia Syndromes. | 6 weeks
  The primary diagnostic endpoint will be determined by the Adjudication Committee using the published criteria for Brugada Syndrome, Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT), Long QT Syndrome (LQTS), Progressive Cardiac Conduction Disease (PCCD), and Short QT Syndrome (SQTS) from the 2013 HRS/EHRA/APHRS Expert Consensus Statement on the Management of Inherited Arrhythmias.
Number of Participants with Adverse Structural and Electrophysiologic Changes to the Atria and Ventricles for Inherited Cardiomyopathy Syndromes. | 6 weeks
  Quantitative imaging and ECG metrics will compare participants who have a pathogenic or likely pathogenic (P/LP) rare variants linked to a CM disease gene compared to controls. Imaging and ECG metrics will be used to assess adverse structural and electrophysiologic changes to the atria and ventricles from inherited cardiomyopathy syndromes. Quantitative metrics will be assessed from contrast-enhanced MRI, signal-averaged ECG, resting 12- lead ECG, Stress treadmill ECG, and ambulatory ECG monitor. Results will be used to test the hypothesis that cases have increased measures of proarrhythmic structural and electrophysiologic changes compared to controls by imaging and ECG endpoints.
Number of Participants with Adverse Structural and Electrophysiologic Changes to the Atria and Ventricles for Inherited Arrhythmia Syndromes. | 6 Weeks
  Quantitative imaging and ECG metrics will compare participants who have a P/LP rare variants linked to an inherited arrhythmia disease gene and will compare to controls. Imaging and ECG metrics will be used to assess adverse structural and electrophysiologic changes to the atria and ventricles from inherited arrhythmia syndromes. Quantitative metrics will be assessed from resting 12- lead ECG, Stress treadmill ECG, and ambulatory ECG monitor. A procainamide challenge will be used on select participants with a non-diagnostic (type II or III) Brugada pattern identified on their previous resting 12-lead ECG or who are P/LP variant carriers in an identified Brugada susceptibility gene. Results will be used to test the hypothesis that cases have increased measures of proarrhythmic structural and electrophysiologic changes compared to controls by imaging and ECG endpoints.
Number of Participants with Changes in Management of Inherited Arrhythmia and CM Syndromes. | 6 weeks
  The Adjudication Committee will determine the management recommendations for each participant at the time of case review. The primary analysis will focus on changes in each management category (e.g., medical therapy, physical activity restrictions, stroke prophylaxis, implantable cardioverter-defibrillator utilization) that resulted from discovery of a rare variant, and a secondary analysis will compare the management in each category regardless of whether it was pre-existing or newly initiated. The participant will be contacted, the results will be reviewed by the principal investigator or coinvestigators to discuss the results of the testing. Any recommendations regarding clinical care will be communicated to the participants existing physicians and ensure adequate follow-up is arranged or will assist the participant in establishing care with a qualified physician.

CONTACTS AND LOCATIONS:
Overall Officials: M. B Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shoemaker MB, Shah RL, Roden DM, Perez MV. How Will Genetics Inform the Clinical Care of Atrial Fibrillation? Circ Res. 2020 Jun 19;127(1):111-127. doi: 10.1161/CIRCRESAHA.120.316365. Epub 2020 Jun 18. PMID 32716712
- [Result] Yoneda ZT, Anderson KC, Quintana JA, O'Neill MJ, Sims RA, Glazer AM, Shaffer CM, Crawford DM, Stricker T, Ye F, Wells Q, Stevenson LW, Michaud GF, Darbar D, Lubitz SA, Ellinor PT, Roden DM, Shoemaker MB. Early-Onset Atrial Fibrillation and the Prevalence of Rare Variants in Cardiomyopathy and Arrhythmia Genes. JAMA Cardiol. 2021 Dec 1;6(12):1371-1379. doi: 10.1001/jamacardio.2021.3370. PMID 34495297
- See also: How Will Genetics Inform the Clinical Care of Atrial Fibrillation? — https://pubmed.ncbi.nlm.nih.gov/32716712/
- See also: Early-Onset Atrial Fibrillation and the Prevalence of Rare Variants in Cardiomyopathy and Arrhythmia Genes — https://pubmed.ncbi.nlm.nih.gov/34495297/

DOCUMENTS (1):
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT05190679/ICF_002.pdf